CLINICAL TRIAL: NCT04607317
Title: A Telehealth Physical Exercise Intervention for the Treatment of Drug Resistant Epilepsy
Brief Title: Exercise as Adjunctive Treatment for Refractory Epilepsy
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: did not enroll as many as planned
Sponsor: Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: IRB00068408
Record Dates: First submitted 2020-10-23; First posted 2020-10-29 (Actual); Last update posted 2022-12-07 (Actual); Status verified 2022-02

CONDITIONS: Refractory Epilepsy; Epilepsy
Keywords: exercise; telehealth; adjunctive treatment
MeSH Terms: conditions — Drug Resistant Epilepsy; Epilepsy; Motor Activity | interventions — Resistance Training

STUDY DESIGN:
Intervention Model Description: Subjects will be randomized to exercise intervention arm or control arm.
Who Masked: Care Provider, Investigator, Outcomes Assessor
Masking Description: Due to the nature of the intervention, participants will not be blinded as to whether they are in the intervention or control group.
  Blinded study staff will perform all pre-and post outcome assessments. The PI will also be blinded
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exercise Intervention (Experimental): Participants in this arm will be enrolled in a telehealth-delivered exercise program with the goal of progressing to 150 min/week (5 days per week, 30 minutes of steady state walking per day). Participants will meet weekly 1:1 with a trained health coach via a Webex platform. Weekly exercise goals will be tailored to the individual's abilities and specific barriers. Coaching will utilize social cognitive theory and self-determination theory to develop self-efficacy for sustainable behavior change.
  Interventions: Behavioral: Exercise program; Behavioral: Health Coach
- Control (Active Comparator): Participants randomized to the wait-list attention control group will continue to undergo standard care for 12 weeks. They will continue to wear the Garmin activity tracker and can view their activity but will not be given an exercise program. They will be contacted by a study coordinator via telephone every 2 weeks for health education. During this time, they will review resources and healthy lifestyle guidelines for people with epilepsy, including healthy diet, medication compliance, seizure precautions, stress management, and sleep hygiene.
  Interventions: Behavioral: Health Information

INTERVENTIONS:
Behavioral: Exercise program — a telehealth-delivered exercise program with the goal of progressing to 150 min/week (5 days per week, 30 minutes of steady state walking per day)
  Arms: Exercise Intervention
Behavioral: Health Coach — The coach will work directly with each participant during their once-weekly virtual 1:1 meeting to progress intensity and duration. Participants will meet with the coach to review a brief social cognitive theory-based module, which will provide education on core behavior change concepts and the benefits of physical activity for those with epilepsy. The coach will review the previous week's exercise during meetings, and will then work with the participant to revise and reset goals for the coming week.
  Arms: Exercise Intervention
Behavioral: Health Information — Participants will be contacted by a study coordinator via telephone every 2 weeks for health education. During this time, they will review resources and healthy lifestyle guidelines for people with epilepsy, including healthy diet, medication compliance, seizure precautions, stress management, and sleep hygiene.
  Arms: Control

SUMMARY:
The purpose of this research study is to determine whether a 12-week telehealth aerobic exercise intervention is feasible in people with epilepsy.

The study team will also gather information on the effect of the intervention on sleep and stress as mediators of seizure frequency, well as effects on epilepsy and epilepsy associated comorbidities.

DETAILED DESCRIPTION:
This is a randomized, controlled pilot trial to assess the feasibility and fidelity of a 12 week, individualized, telehealth exercise intervention in people with refractory epilepsy. This will be carried out using a 2 arm, parallel group design with a waitlist attention control.

Participants will undergo formal exercise testing prior to enrollment to determine safety and establish a baseline fitness level. Participants will use a wrist-worn Garmin device to record activity and sleep. After a 4 week baseline period, participants will be randomized to intervention or wait-list attention control. The intervention group will undergo a 12-week telehealth exercise program designed by a trained health coach and tailored to the individual's personal fitness level and exercise preferences. The intervention is based in social cognitive theory to implement and enforce sustainable behavior change. The wait-list attention control will receive health education but will not be given an exercise program. At the end of the intervention period, the control group will be given the option to participate in the exercise program.

The study will assess recruitment and retention as well as fidelity, acceptability and sustainability of a telehealth exercise intervention in this population.

The study will investigate objective and subjective measures of the effect of the intervention on the known seizure triggers of sleep and stress as possible mediators of seizure frequency.

The study will collect information regarding the effects of the intervention on depression, anxiety, quality of life, cognition, and seizure frequency.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 or older
* Focal or generalized epilepsy, as clinically determined by a Wake Forest Baptist Health epileptologist.
* Seizure frequency of at least 1 clinically observable seizure in the year prior to enrollment
* Able to ambulate independently without assistive device
* Access to a smartphone with application capabilities
* Internet access or cellular data plan to attend virtual sessions

Exclusion Criteria:

* Diagnosis of nonepileptic or psychogenic spells
* Seizures associated with frequent falls with injury
* <50% adherence with wearing the device or completing the study diary during the baseline period.
* Currently in an exercise program
* Medical conditions that would limit ability to participate in an exercise intervention such as:
* Stage III or IV Congestive Heart Failure (CHF)
* End-stage Renal Disease
* Severe dementia or significant cognitive impairment
* Uncontrolled hypertension (HTN)
* Motor conditions that limit ambulation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2021-04-13 (Actual); Primary Completion 2022-05-31 (Actual); Study Completion 2022-05-31 (Actual)

PRIMARY OUTCOMES:
Proportion of participants recruited | Week 0 Baseline
  This outcome measure assesses Feasibility of Recruitment. Recruitment will be calculated as a percentage by dividing the total number of enrolled participants by the total number of eligible participants.
Proportion of participants completing all visits | Visit 3 (Week 16 after Baseline)
  This outcome measure assesses Feasibility of Retention. Retention will be calculated as the percentage of all participants who complete Visit 2 Week 16 (End of Intervention) out of the total number of participants enrolled.

SECONDARY OUTCOMES:
Proportion of Participants who achieve their target | Visit 3 (Week 16 after Baseline)
  Fidelity of the Intervention is the proportion of participants in the intervention group who achieve their target HR for at least 80% of their individually prescribed weekly minutes. A priori goal 70% of participants achieve this in at least 10 out of the 12 weeks of the intervention
Acceptability of the Intervention Questionnaire | Week 16 and Week 28 after baseline
  This will be a qualitative measure based on post program question of how satisfied the subject was with the exercise intervention with a scale of 1=Very Unsatisfied, 2=Unsatisfied, 3=Neutral, 4=Satisfied, 5=Very Satisfied. Results will include percentage of people who answer 4 or above.
Percentage of participants achieving the goal for at least 10 weeks | Week 28 after baseline
  Sustainability of the intervention is defined as maintenance of at least 80% of the last assigned weekly minutes in target HR zone each week. The intervention will be considered sustainable if 60% of the participants achieve this goal for at least 10 out of the 12 follow-up weeks.

OTHER OUTCOMES:
Heart Rate Variability (HRV) measurement | baseline and Visit 3 (week 16 after baseline)
  Continuous heart rate will be recorded while the participant is breathing normally in seated position for 10 minutes. This will be assessed by sympathetic and parasympathetic activity expressed as low-frequency (LF) and high-frequency (HF) power spectrum, standard deviation of NN intervals (SDNN), and the root mean square of successive differences (RMSSD).
Perceived Stress Scale (PSS) | baseline, week 16 after baseline, week 28 after baseline
  A validated measure of the subjective stress experience which has been shown to correlate with systemic stress hormones. Individual scores can range from 0 to 40 with higher score indicating higher perceived stress. Scores ranging from 0-13 would be considered low stress.
Pittsburgh Sleep Quality Index (PSQI) | baseline, week 16 after baseline, week 28 after baseline
  Scores range from 0-21 with higher score indicating worse sleep quality. A common cutoff for poor sleep quality is score greater than 5.
Nightly average total sleep time (TST) | baseline, week 16 after baseline, week 28 after baseline
  will be collected from the wearable device
Change in Seizure Frequency | baseline, week 16 after baseline, week 28 after baseline
  the number of seizures during the final 4 weeks of the intervention will be compared to the number of seizures during the 4 week baseline.
Neurological Disorders Depression Inventory for Epilepsy (NDDI-E) | baseline, Visit 3 (week 16 after baseline)
  Scores range from 6-24 with higher scores indicating higher risk for depression. A common cutoff is that a score greater than 15 is suggestive of major depression.
Generalized Anxiety Disorder (GAD-7) | baseline, week 16 after baseline, week 28 after baseline
  Scores range from 0-21. A score of 10 or greater suggests high risk for Generalized Anxiety Disorder (GAD), while scores of 5-9, 10-14, and 15-21 could represent mild, moderate, and severe GAD.
Test of Premorbid Functioning (TOPF) | baseline
  TOPF is a test of static cognitive function. This is a standard score with a mean of 100 and a standard deviation of 15. The score can range from ~60-145. This is a single word reading test that is used to estimate premorbid functioning. A higher score denotes a better outcome.
Wechsler Adult Intelligence Scale - 4th edition (WAIS-IV) | baseline and week 16 after baseline
  Digit Span Subtest. A common measure of current overall intellectual functioning. This scale produces a standard score with a mean of 100 and a standard deviation of 15. A higher score is better.
Controlled Oral Word Association Test (COWAT) | baseline and week 16 after baseline
  This test produces a T score with a mean of 50 and an standard deviation of 10. It measures lexical and semantic verbal fluency.
Rey Auditory Verbal Learning Test (RAVLT) | baseline and week 16 after baseline
  This test produces a T score with a mean of 50 and a standard deviation of 10. It measures verbal learning and memory.
Delis-Kaplan Executive Function Stroop Test | baseline and week 16 after baseline
  This test produces a scaled score of 10 with a standard deviation of 3. It measures cognitive inhibition.
Physical Function: walk test | baseline and week 16 after baseline
  Measure of cardiorespiratory fitness. Distance walked in 6 minutes.
Quality of Life in Epilepsy-31 (QOLIE-31) | baseline, week 16 after baseline, week 28 after baseline
  Score ranges from 0-100 with higher score indicating better quality of life.
Exercise Self-Efficacy Questionnaire (EXSE) | baseline, week 16 after baseline, week 28 after baseline
  Items on all self-efficacy questionnaire that ask participants to rate their confidence on a 100-point percentage scale such that 0% corresponds with "not confident at all", and 100% corresponds with "highly confident", and scale scores are generated by averaging all items in the scale. Higher scores represent greater self-efficacy.
Exercise Goal Setting Questionnaire (EGS) | baseline, week 16 after baseline, week 28 after baseline
  This questionnaire assesses participants' ability to set and meet goals relative to exercise behavior by asking how closely a series of statements describes them (e.g., "I usually set dates for achieving my goals") on a 5 point scale such that 1 corresponds with "Does not Describe" and 5 corresponds with "Describes Completely". A total scale score was generated by summing all items, with possible scores ranging from 10 to 50 with higher scores reflecting greater goal setting behavior
Multidimensional Expectations for Exercise Scale (MOEES) Physical Score | baseline, week 16 after baseline, week 28 after baseline
  This 15-item questionnaire assesses the three dimensions of outcome expectations for exercise (i.e., physical, social, and self-evaluative). Participants are asked to rate the degree to which they agree with statements relating to outcome expectations (e.g., "Exercise will increase my muscle strength") on a 5-point scale. Three subscale scores will be generated. Physical scores range from 6 to 30 with higher scores indicating higher levels of outcome expectations for exercise.

CONTACTS AND LOCATIONS:
Overall Officials: Halley Alexander, MD, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Wake Forest University Health Sciences, Winston-Salem, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Informed Consent Form (2022-04-05): https://cdn.clinicaltrials.gov/large-docs/17/NCT04607317/ICF_000.pdf